CLINICAL TRIAL: NCT00469872
Title: Family Centred Functional Therapy for Children With Cerebral Palsy
Brief Title: Focus on Function Study for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Mary Law, Professor, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD044444 (NIH)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child Focused (Active Comparator): Occupational and physical therapy focused on improving child's skills and abilities through rehabilitation to improve child functioning
  Interventions: Procedure: Context-focused compared to child-focused interventions
- Context Focused (Experimental): Occupational and physical therapy focused on improving child's skills and abilities through rehabilitation to change the task or environment around a child
  Interventions: Procedure: Context-focused compared to child-focused interventions

INTERVENTIONS:
Procedure: Context-focused compared to child-focused interventions

SUMMARY:
This study will compare two treatment approaches that are currently being used for children with cerebral palsy. Both treatments aim to improve a child's function. The two approaches being compared are: 1) improving function by working with the child to improve his/her skills and abilities ("child-focused" approach) and 2) improving function by changing/adapting the task and/or environment around the child to improve his/her skills and abilities ("context-focused" approach). It is hypothesized that the context-focused approach will significantly improve activity and participation outcomes while leading to no significant decreases in body function and structure outcomes.

DETAILED DESCRIPTION:
Children with cerebral palsy commonly receive ongoing physical and occupational therapy to facilitate development and to enhance functional independence in movement, self-care, play, school activities and leisure. The primary objective of this project is to conduct a multi-site clinical trial to evaluate the efficacy of a context-focused approach in improving performance of functional tasks, mobility, participation in everyday activities and quality of life in 220 children 12 months to 5 years of age who have cerebral palsy. A randomized clinical trial research design will be used to examine the efficacy of the context-focused approach compared to a child-focused approach. 72 therapists in Ontario and Alberta will be randomly assigned to provide either context-focused or child-focused therapy. Therapists in both groups will participate in a training workshop and expert consultants will be available to support the therapists throughout the study. Children will receive either the context-focused or child-focused therapy intervention for a period of 6 months. Outcomes will be evaluated at baseline, after 6 months of treatment and at a 3-month follow-up period. Outcomes will be measured across the domains of the International Classification of Functioning, Disability and Health, including body function and structure (range of motion, spinal alignment), activities (performance of functional tasks, motor function), participation (involvement in formal and informal activities), and environment (parent perceptions of care, parental empowerment). The children's range of motion will also be evaluated by an independent, trained evaluator at baseline, 3, 6, and 9 months. We hypothesize that the context-focused approach will significantly improve activity and participation outcomes while leading to no significant decreases in body function and structure outcomes.

ELIGIBILITY:
Inclusion Criteria:

* children with cerebral palsy
* children classified as levels I-V on the Gross Motor Function Classification System
* children aged 12 months to 5 years, 11 months

Exclusion Criteria:

* children whose parents feel uncomfortable or unable to respond to interviews and questionnaires in English
* children with planned surgical or medication changes during the study period that may impact motor function
* parents and caregivers who state that they will not be able to comply with the treatment schedule

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
activities (performance of functional tasks, motor function) | 6 months

SECONDARY OUTCOMES:
body function and structure (range of motion) | 6 months
particpation | 6 months
parental empowerment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Law, PhD, Principal Investigator — McMaster University; Johanna Darrah, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - McMaster University, Hamilton, Ontario

REFERENCES:
- [Derived] Law M, Darrah J, Pollock N, Rosenbaum P, Russell D, Walter SD, Petrenchik T, Wilson B, Wright V. Focus on Function - a randomized controlled trial comparing two rehabilitation interventions for young children with cerebral palsy. BMC Pediatr. 2007 Sep 27;7:31. doi: 10.1186/1471-2431-7-31. PMID 17900362